CLINICAL TRIAL: NCT04284696
Title: Chewing Gum Containing Vitamin-c to Treat Emesis Gravidarum: a Randomized Controlled Trial
Brief Title: Chewing Gum Containing Vitamin-c to Treat Emesis Gravidarum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alex Farr, MD PhD, Assistant Professor, Consultant Physician, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1949-2019
Record Dates: First submitted 2019-10-20; First posted 2020-02-26 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hyperemesis Gravidarum; Nausea Gravidarum; Vitamin C Deficiency
MeSH Terms: conditions — Hyperemesis Gravidarum; Ascorbic Acid Deficiency | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum (Active Comparator): patients with emesis gravidarum who take a chewing gum with vitamin C (verum) "ad libitum" several times daily for 2 weeks
  Interventions: Dietary Supplement: Pregnan-C-Gum(R) chewing gum
- Placebo (Placebo Comparator): patients with emesis gravidarum who take chewing gum without vitamin C (placebo) "ad libitum" several times daily for 2 weeks
  Interventions: Dietary Supplement: Placebo chewing gum
- Nihil (No Intervention): patients with emesis gravidarum who do not use chewing gum during the study phase

INTERVENTIONS:
Dietary Supplement: Pregnan-C-Gum(R) chewing gum — Using a chewing gum with 150mg vitamin C (per piece/gum) for 14 days "ad libitum"
  Arms: Verum
Dietary Supplement: Placebo chewing gum — Using a chewing gum without vitamin C (per piece/gum) for 14 days "ad libitum"
  Arms: Placebo

SUMMARY:
Nausea and vomiting is a common complication of pregnancy and occurs in 70-80% of all pregnancies. The symptoms usually start 2-4 weeks after fertilization and peak between the 9th and 16th week of gestation. In the 22nd week of pregnancy, the symptoms usually resolve. In up to 10% of all pregnancies nausea and vomiting may persist until delivery, which is called emesis gravidarum. In 0.3-2% of all pregnancies, nausea and vomiting occur with a pathological intensity called hyperemesis gravidarum. The cause of nausea and vomiting during pregnancy is unknown, but it is believed that the stimulus is the placenta and not the fetus. Antihistamines have proven to be an effective therapy. Histamine is increasingly produced during pregnancy by mast cells in the endometrium and myometrium, but also by mast cells in the placenta and in the decidua. High expression of the histamine-producing enzyme histamine-decarboxylase (HDC) in the placenta and many histamine receptors at the feto-maternal transition in the decidua indicate a physiological role of the histamine during pregnancy. The antidote is diamine oxidase (DAO), which is produced in the decidua and trophoblast and breaks down histamine. DAO acts as a barrier to prevent excessive passage of histamine into the maternal and fetal circulation. DAO levels increase exponentially in the first 20 weeks of pregnancy to 1000 times the baseline before pregnancy. It has been shown that intravenous vitamin C significantly reduces blood histamine levels in both allergic and non-allergic disorders. Another study with the German Navy also proved that oral vitamin C administration can reduce nausea in seasickness. In an Australian study in 2016, it was shown that chewing gum was not inferior to ondansetron therapy in patients with postoperative nausea and vomiting (PONV). From the available literature, we conclude that high maternal histamine concentrations in early pregnancy may be a cause of nausea and vomiting, whereas DAO is not sufficiently expressed by the transfer of histamine from the decidua and trophoblast into the maternal circulation prevent. Vitamin C has been identified in controlled clinical trials as a way to lower blood histamine levels. Furthermore, chewing gum was already described as a treatment option for nausea and vomiting. The aim of this study is therefore to test whether chewing gum containing vitamin C in pregnant women with emesis gravidarum has the potential to reduce nausea and vomiting and to evaluate a possible association between maternal human chorionic gonadotropin (hCG) or histamine levels and the severity of nausea and vomiting in early pregnancy as well as the influence of other factors such as thyroxine and pyridoxine.

DETAILED DESCRIPTION:
The following 3 groups of patients should be compared: (1) patients with emesis gravidarum who take a chewing gum with vitamin C (verum) "ad libitum" several times daily for 2 weeks; (2.) patients with emesis gravidarum who take chewing gum without vitamin C (placebo) "ad libitum" several times daily for 2 weeks; (3.) patients with emesis gravidarum who do not use chewing gum during the study phase. The enrollment will take place at the Department of Obstetrics and Gynecology, Division of Obstetrics and Feto-Maternal Medicine, at the Medical University of Vienna. All pregnant women in the first trimester, who present for triage and birth registration between 6 to 9 gestational weeks, complaining of nausea and meeting the inclusion criteria, will be offered to participate in the study. If they agree to participate, patients will be randomized to one of the 3 study groups. In case of enrollment, patients are not allowed to take any other nausea therapy during the study period, otherwise the results could be distorted. Both the vitamin C-containing chewing gums (verum) and the non-vitamin C-containing chewing gums (placebo) are manufactured by the company Frey AG (Migros-Genossenschafts-Bund, 8031 Zurich, CH). Both chewing gums are not distinguishable from each other in taste. The only difference between verum and placebo is the proportion of 150mg vitamin C per chewing gum (for verum) or no vitamin C (for placebo). The other ingredients are as follows: sweeteners isomalt, sorbitol, maltisirup, sucralose, acesulfame K, chewing gum (with antioxidant E306), sodium L-ascorbate, flavorings, acidifier (apple and citric acid), thickener gum arabic, dye E171, humectant E422 and E1518, coating agents E903 and E553b. The randomization takes place by means of the GCP-compliant web-based randomizer of the Institute of Medical Informatics, Statistics and Documentation (IMI) of the Medical University of Graz (license Meduni Vienna). The ratio of the allocation to the 3 groups is 1:1:1. Furthermore, as co-variable nicotine abuse is included in the randomization, since smoking with a lower risk correlates with suffering from hyperemesis gravidarum. Study patients are asked to complete a validated questionnaire (modified PUQE-Score) on their condition. In addition, there is a blood sampling for the determination of human chorionic gonadotropin (hCG), diamine oxidase (DAO), thyroxine, pyridoxine and the histamine concentration in the blood of the patient. Patients are subsequently evaluated at two further follow-up appointments, one in the course of routine retesting for cervical crease measurement (between 11-14 weeks of gestation) and 2nd time during routine organ screening (between 20-24 weeks of gestation). At these appointments, the same blood sampling is repeated and the evaluation of well-being using the Modified PUQE questionnaire are carried out again. With the second control appointment the supervision ends within the study. The study phase is thus completed at the latest at the time of the organ screening at the Department of Obstetrics and Gynecology, at the latest until the 24th week of pregnancy. For the determination of DAO, hCG, thyroxine, pyridoxine and histamine, the following tubes (a total of 32mL blood) are necessary: 3 serum tube of 8mL with separating gel (DAO, hCG, thyroxine, pyridoxine) + 1 EDTA tube of 8mL (histamine). In addition, it is planned to store the material that has not been used for the determination of blood concentrations in order to answer future questions in the field of biomedical research in the MedUni Vienna Biobank. The legal basis for this can be found in the Research Organization Act 2018 §2d. For each additional project that uses samples and / or data from this study, a separate report will be sent to the Ethics Committee of the Medical University of Vienna. The analysis of the DAO levels takes place in the Allergy Center Floridsdorf, which has many years of experience in the measurement of DAO and is considered a reliable partner. The samples are pseudonymized and stored at -80°C. The measurement of of the other blood levels is carried out by the Clinical Institute for Laboratory Medicine at the Medical University of Vienna. The samples are taken directly after acceptance by means of a cooled transport container on site for analysis (coordinated preanalytics). The design of the planned study is prospective, randomized, double-blind, placebo-controlled. Blinding is provided between verum and placebo chewing gum (groups 1-2). The taste of verum and placebo chewing gum is identical. The non-inferiority of chewing gum chewing against doing nothing should also be proved. In addition to the course of objective parameters such as DAO, hCG and histamine, the personal condition of the affected patient should be assessed on the basis of the modified PUQE score. The number of ingested chewing gum is determined by means of the number of used packs on the 1st inspection date. In addition, maternal characteristics are collected, which should be descriptive and should be included in the multivariate model: age, pregnancy, parity, gestational age at diagnosis, comorbidities, long-term medication, complications in this or previous pregnancies, previous hyperemesis gravidarum, nicotine abuse, educational level. In addition, the pregnancy outcome is retrospectively assessed in order to evaluate any influence of the chewing gum containing vitamin C on the pregnancy outcome. The primary endpoint is the modified PUQE score for the 1st control appointment. Secondary endpoints are the PUQE score at the 2nd control appointment, as well as DAO and histamine concentrations for the 1st and 2nd control appointment. About the statistical methods: Based on the work of Birkeland E et al., a standard deviation of 3 points or less can be assumed for each Modified PUQE score group. Power analysis was conducted in preparation of the study, thereby a caseload of 111 patients was calculated to find differences between the groups with a power of >80%. Descriptive statistics (number, mean, standard deviation, median, minimum and maximum) should be given separately for the 3 target variables Modified PUQE score, DAO and histamine values for the 3 measurement times. The data is also displayed graphically using box plots and trajectories. Further metric variables are also described by mean, standard deviation, median, minimum and maximum, categorical variables are described by absolute and relative frequencies. As a primary analysis, a mean value comparison of the Modified PUQE scores is performed between the 3 groups for the measurements at the 2nd control date. For this, an ANCOVA model is calculated, to which the respective initial values at birth registration and the week in which the second measurement takes place are considered as covariates. From the ANCOVA model, the null hypothesis that there are no group differences on average is tested with an F-test at the 5% significance level. If this global null hypothesis is discarded, all pairwise group comparisons are performed by T tests for the corresponding model coefficients of the ANCOVA model at the 5% significance level. This test procedure does not require any further correction for multiple testing when comparing 3 groups. In another exploratory model, the maternal characteristics listed in the preceding section are additionally included as covariates to investigate the potential influence of these variables on the Modified PUQE score and to calculate adjusted group differences. The secondary endpoints are compared to the primary endpoint using ANCOVA models between the three groups. As a further analysis, the Spearman correlations between the Modified PUQE scores, hCG, DAO, thyroxine, pyridoxine and histamine levels at the three different time points will be determined.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* singleton pregnancy
* signed information sheet
* symptoms of nausea and / or vomiting in early pregnancy
* no pre-existing medication for nausea and vomiting

Exclusion criteria:

* age <18 years
* multiple pregnancy
* patients with gastric band or in Z.n. bariatric surgery
* preexisting diabetes mellitus or gestational diabetes
* inability to consent to participation in the study
* already started therapy against the emesis gravidarum
* taking any antiemetic drugs during the study phase

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Enrollment: 126 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Modified PUQE (Pregnancy-Unique Quantification of Emesis and Nausea) Score | 1 month
  validated questionnaire describing individual nausea

SECONDARY OUTCOMES:
Level of diamine oxidase (DAO) serum concentratlon | 1 month
  maybe an antidot of nausea and vomiting
Level of histamine serum concentration | 1 month
  maybe a cause of nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Alex Farr, MD PhD, Principal Investigator — Medical University of Vienna, Department of Obstetrics and Gynecology; Vienna General Hospital
Locations (1):
- Medical University of Vienna, Dept. of Obstetrics and Gynecology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No